CLINICAL TRIAL: NCT00586599
Title: Levels of the Stat4 Alpha and Stat4 Beta Isoforms in PBMCs From Patients With Crohn's Disease and Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0707-69; IRB # 0707-69
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: IBD; CD; UC; Crohn's Disease; Ulcerative Colitis; Pediatric; inflammatory markers
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Other): Subjects who have no inflammatory disease who will be age/gender matched controls for the 2 other arms.
  Interventions: Other: measurement of inflammatory markers
- IBD and infliximab (Other): Subjects who have IBD and will be receiving infliximab for the first time.
  Interventions: Other: measurement of inflammatory markers
- Newly Diagnosed IBD (Other): Subjects who are newly diagnosed with IBD and given corticosteroid therapy.
  Interventions: Other: measurement of inflammatory markers

INTERVENTIONS:
Other: measurement of inflammatory markers — measuring inflammatory markers and comparing to controls.

SUMMARY:
The goal in these studies will be to assess the relative levels of the Stat4 alpha and Stat4 beta isoforms in PBMCs from patients with Crohn's Disease, ulcerative colitis, celiac disease or from control patients. We hypothesize that the beta to alpha ratio will be higher in patients with active disease and that there will be a correlation between the ratio and the severity of disease.

ELIGIBILITY:
Inclusion Criteria:

* Children with a new diagnosis of Crohn's Disease and whose physician has not yet initiated corticosteroid treatment (10 Subjects):
* Clinical diagnosis within the previous 21 days
* Above age 7 and younger than age 18
* Signed informed consent statement and assent statement.
* Children with a new diagnosis of Ulcerative Colitis and whose physician has not yet initiated corticosteroid treatment (10 Subjects):
* Clinical diagnosis within the previous 21 days
* Above age 7 and younger than age 18
* Signed informed consent statement and assent statement.
* Children with Crohn's Disease whose physician has initiated Infliximab treatment for the first time (10 Subjects):
* Clinical diagnosis of Crohn's Disease
* Above age 7 and younger that age 18
* Signed informed consent statement and assent statement.
* Children with Ulcerative Colitis whose physician has initiated Infliximab treatment for the first time (10 Subjects):
* Clinical diagnosis of Ulcerative Colitis
* Above age 7 and younger than age 18
* Signed informed consent statement and assent statement.
* Healthy Controls (10 Subjects):
* Above age 7 and younger than age 18
* otherwise healthy, with no intercurrent illness as determined by a member of the study team using the eligibility checklist
* controls will be gender and age (± 2 years) matched to the patient groups described above
* Signed informed consent statement and assent statement

Exclusion Criteria:

* unwilling to give consent for this study.
* child with prior prescription and administration of Infliximab

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2007-08; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
This study hopes to assess the relative levels of the Stat4a and Stat4β isoforms in PBMCs from patients with Crohn's Disease, ulcerative colitis, or from control patients. | Total duration of treatment will be 20-24 weeks (Arm A and Arm B) or 50-54 weeks (Arm C/ Arm D).

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Steiner, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University-Riley Hospital, Indianapolis, Indiana, United States